CLINICAL TRIAL: NCT02584959
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Two-period, Three-sequence, Partial Crossover Study to Evaluate the Efficacy and Safety of Subcutaneous Administration of 2000 IU of C1 Esterase Inhibitor [Human] Liquid for Injection for the Prevention of Angioedema Attacks in Adolescents and Adults With Hereditary Angioedema
Brief Title: Study to Evaluate the Clinical Efficacy and Safety of Subcutaneously Administered C1 Esterase Inhibitor for the Prevention of Angioedema Attacks in Adolescents and Adults With Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SHP616-300
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Experimental/Placebo (Experimental): Subjects will be randomized to receive C1 Esterase Inhibitor in the 1st Treatment period and then switch to Placebo in the 2nd treatment period.
  Interventions: Drug: C1 esterase inhibitor [human] liquid; Drug: Placebo
- Placebo/Experimental (Experimental): Subjects will be randomized to receive a placebo treatment in the 1st Treatment period and then switch to receive C1 Esterase Inhibitor in the 2nd treatment period.
  Interventions: Drug: C1 esterase inhibitor [human] liquid; Drug: Placebo
- Experimental/ Experimental (Experimental): Subjects will be randomized and receive C1 Esterase Inhibitor in both 1st as well as the 2nd treatment period
  Interventions: Drug: C1 esterase inhibitor [human] liquid

INTERVENTIONS:
Drug: C1 esterase inhibitor [human] liquid — C1 Esterase Inhibitor [Human] Liquid administered Subcutaneously as specified on specified days
Drug: Placebo — Placebo
  Arms: Experimental/Placebo; Placebo/Experimental

SUMMARY:
The purpose of this study is to assess the efficacy and safety of subcutaneous administration of a liquid formulation of C1 esterase inhibitor for the prevention of angioedema attacks in adolescent and adult subjects with hereditary angioedema.

ELIGIBILITY:
The maximum duration of participation is approximately 9 months. Patients will complete a screening period of up to 21 days. Following screening, eligible patients will be randomly assigned to 1 of 3 treatment sequences. Each patient will undergo 2 14-week treatment periods for a total of 28 weeks (Treatment Period 1 and Treatment Period 2). After completing the 2 treatment periods, patients will enter a 1-month follow-up period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (27):
- United States (16):
  - Medical Research of Arizona, Scottsdale, Arizona
  - AIRE Medical of Los Angeles, Santa Monica, California
  - Bay Area Allergy, Walnut Creek, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Asthma and Allergy Associates PC, Colorado Springs, Colorado
  - Atlanta Allergy and Asthma Clinic, Marietta, Georgia
  - Institute For Asthma and Allergy, Chevy Chase, Maryland
  - Washington University, St Louis, Missouri
  - Allergy Asthma and Immunology, Fair Lawn, New Jersey
  - Allergy Treatment Center of New Jersey, Iselin, New Jersey
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Bernstein Clinical Research Center Inc, Cincinnati, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Allergy Clinic of Tulsa, Tulsa, Oklahoma
  - AARA Research Center, Dallas, Texas
  - Premier Clinical Research, Spokane, Washington
- Canada (2):
  - McMaster University Medical Center, Hamilton, Ontario
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
- Hämophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf, Germany
- Semmelweis Egyetem, Budapest, Hungary
- Israel (2):
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- MediQuest Clinical Research Center, Târgu Mureş, Romania
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Lumry WR, Martinez-Saguer I, Yang WH, Bernstein JA, Jacobs J, Moldovan D, Riedl MA, Johnston DT, Li HH, Tang Y, Schranz J, Lu P, Vardi M, Farkas H; SAHARA study group. Fixed-Dose Subcutaneous C1-Inhibitor Liquid for Prophylactic Treatment of C1-INH-HAE: SAHARA Randomized Study. J Allergy Clin Immunol Pract. 2019 May-Jun;7(5):1610-1618.e4. doi: 10.1016/j.jaip.2019.01.021. Epub 2019 Jan 23. PMID 30682573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 33 sites/centers in 7 countries: United States, Canada , Germany, Hungary, Israel, Spain, and Romania .
Pre-assignment Details: Of the 81 participants screened, 6 subjects failed to meet the randomization criteria and were not randomly assigned to a treatment sequence . All 75 randomly assigned participants received at least 1 dose of the IP.
Groups:
- Experimental/Placebo: Participants were randomized to receive C1 Esterase Inhibitor in the 1st treatment period and then switched to Placebo in the 2nd treatment period.
- Placebo/Experimental: Participants were randomized to receive placebo treatment in the 1st treatment period and then switched to receive C1 Esterase Inhibitor in the 2nd treatment period.
- Experimental/ Experimental: Participants were randomized to receive C1 Esterase Inhibitor in both 1st as well as the 2nd treatment period.
Period: Period 1
Arm/Group | Experimental/Placebo | Placebo/Experimental | Experimental/ Experimental
Started | 31 | 29 | 15
Completed | 28 | 25 | 15
Not Completed | 3 | 4 | 0
Not completed — Withdrawn from study | 3 | 4 | 0
Period: Period 2
Arm/Group | Experimental/Placebo | Placebo/Experimental | Experimental/ Experimental
Started | 28 | 25 | 15
Completed | 22 | 24 | 13
Not Completed | 6 | 1 | 2
Not completed — Withdrawn from study | 6 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental/Placebo | Placebo/Experimental | Experimental/ Experimental | Total
Number analyzed (Participants) | 31 | 29 | 15 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 1 | 3
  Between 18 and 65 years | 30 | 25 | 13 | 68
  >=65 years | 1 | 2 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (13.16) | 40.7 (15.34) | 44.4 (16.40) | 41.3 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 8 | 52
  Male | 8 | 8 | 7 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 30 | 27 | 15 | 72
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time-Normalized Number of Attacks (NNA) for Participants During a Treatment Period
Description: The angioedema attacks were recorded in the electronic patient diary. The investigator completed a separate angioedema eCRF for each attack based on the review of the patients diary. Time-normalized number of angioedema attacks was expressed as the number of attacks per month (ie, 30.4 days) of exposure. NNA=30.4 * (number of attacks during treatment period) / (days of treatment period).
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Population: Data were not collected for the Experimental/Experimental Arm for this outcome measure and this represents the full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of attacks
Groups:
- Treatment C1 INH: Participants who received C1 Esterase Inhibitor (C1 INH) treatment (in period 1 of the Experimental/Placebo arm and in period 2 of the Placebo/Experimental arm).
- Treatment Placebo: Participants who received Placebo treatment (in period 2 of the Experimental/Placebo arm and in period 1 of the Placebo/Experimental arm).
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 56 | 57
Number of attacks | 1.611 [1.067 to 2.156] | 3.931 [3.391 to 4.471]
Statistical Analysis 1: Comparison: Treatment C1 INH vs Treatment Placebo; The LS means, 95% CIs, and p-values were based on a mixed effect linear model with period, sequence ,use of prophylactic therapy with C1 INH at randomization, and treatment as fixed effects and subject nested within sequence as a random effect; Test type: Other; p < 0.0001, Mixed Models Analysis; Difference in LS means = -2.320, 95% CI 2-sided [-2.895 to -1.744]

2. Secondary Outcome: Proportion of Participants Meeting at Least a 50% Reduction in NNA (Normalized Number of Angioedema Attacks) During the Experimental Injection Treatment Period Relative to the Placebo Period.
Description: The angioedema attacks were recorded in the electronic patient diary. The investigator completed a separate angioedema eCRF for each attack based on the review of the patients diary. Time-Normalized Number of Attacks was expressed as the number of attacks per month (ie, 30.4 days) of exposure. NNA = 30.4 x (number of attacks during treatment period) / (days of treatment period).
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Population: Analysis done on participants from the crossover sequences (Experimental/Placebo, Placebo/Experimental) who were dosed in both treatment periods. As the measure is implicitly a within subject comparison of the two arms the full analysis set is reported here. Participants with 0 attacks in the placebo period were excluded as %-reduct. not calculated
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Set: Including all participants in the cross-over sequences who had data in both treatment periods and who received at least one dose of C1 Esterase Inhibitor and had at least 1 post-baseline primary efficacy assessment.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 49
Participants | 38

3. Secondary Outcome: Time-Normalized Number of Attacks (NNA) for Participants During Each Treatment Period Excluding the First 2 Weeks.
Description: as for outcome 1
Time Frame: Weeks 3 to 14 for treatment period 1 and 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of Attacks
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 55 | 55
Number of Attacks | 1.524 [0.912 to 2.136] | 3.847 [3.237 to 4.457]
Statistical Analysis 1: Comparison: Treatment C1 INH vs Treatment Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Mixed Models Analysis; Difference in LS means = -2.323, 95% CI 2-sided [-2.969 to -1.677]

4. Secondary Outcome: Proportion of Participants Meeting at Least a 50% Reduction in NNA (Normalized Number of Angioedema Attacks) During the Experimental Injection Treatment Period Relative to the Placebo Period Excluding the First 2 Weeks of Each Treatment Period.
Description: as for outcome 2
Time Frame: Weeks 3 to 14 for treatment period 1 and 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Data Set: Including all participants in the cross-over sequences who had data in both treatment periods and who received at least one dose of C1 Esterase Inhibitor and had at least 1 post-baseline primary efficacy assessment.
Arm/Group | Full Analysis Data Set
Number analyzed (Participants) | 47
Participants | 36

5. Secondary Outcome: Proportion of Participants Meeting at Least a 50% Reduction in NNA (Normalized Number of Angioedema Attacks) During the Experimental Injection Treatment Period Relative to the Pre-treatment Assessment.
Description: as for outcome 2
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Population: Full analysis set from the crossover sequences (Experimental/Placebo arm and Placebo/Experimental arm) was used for analysis of this outcome measure.Participants with zero attacks in the placebo period were excluded because a percent reduction could not be calculated. Analysis was done on participants with pretreatment and post-treatment NNA values
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 53 | 55
Participants | 41 | 13

6. Secondary Outcome: Cumulative Attack Severity
Description: Severity of the angioedema attack sign/symptom was characterized as None: no symptom; Mild: noticeable symptom but easily tolerated by the participant and did not interfere with routine activities; Moderate: symptom interfered with the participant's ability to attend school or participate in family life and social/recreational activities; Severe: symptom significantly limited the participant's ability to attend school or participate in family life and social/recreational activities. Symptom severity score was assigned as Mild = 1, Moderate = 2 and Severe = 3. Cumulative attack severity score was the sum of the maximum symptom severity scores recorded for each angioedema attack in a treatment period. Cumulative attack-severity score normalized per month [(raw score/number of days of participation in that treatment period)*30.4] was reported here. Cumulative attack-severity score normalized per month ranged from 0 to 19.83 and higher scores represent worse symptoms.
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 56 | 57
Score on a scale | 3.159 [1.856 to 4.463] | 8.041 [6.746 to 9.336]
Statistical Analysis 1: Comparison: Treatment C1 INH vs Treatment Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Mixed Models Analysis; Difference in LS means = -4.881, 95% CI 2-sided [-6.113 to -3.649]

7. Secondary Outcome: Number of Attack-free Days
Description: Attack free days were normalized per month.
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 56 | 57
Days | 26.788 [25.106 to 28.470] | 21.353 [19.681 to 23.025]
Statistical Analysis 1: Comparison: Treatment C1 INH vs Treatment Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; Difference in LS means = 5.435, 95% CI 2-sided [3.981 to 6.889]

8. Secondary Outcome: Number of Angioedema Attacks Requiring Acute Treatment
Description: Angioedema attacks were normalized per month.
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of attacks
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 56 | 57
Number of attacks | 1.454 [0.906 to 2.002] | 3.628 [3.085 to 4.172]
Statistical Analysis 1: Comparison: Treatment C1 INH vs Treatment Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; Difference in LS means = -2.175, 95% CI 2-sided [-2.750 to -1.599]

9. Secondary Outcome: Response to Icatibant When Administered for an Acute Attack
Description: The number of Acute Hereditary Angioedema Attacks that required Icatibant as acute therapy is presented by the number of Icatibant injections.
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Population: For treatment with C1 INH (Overall treatment with C1 INH group) all participants who received C1 INH in each of the randomized arms (experimental/placebo, placebo/experimental and experimental/experimental) are included.
Measure: Count of Units; unit: Attacks requiring Icatibant
Units Other Than Participants: Attacks requiring Icatibant
Groups:
- Treatment C1 INH: Participants who received C1 Esterase Inhibitor (C1 INH) treatment (in period 1 of the Experimental/Placebo arm, in period 2 of the Placebo/Experimental arm and in period 1 and 2 of the Experimental/Experimental arm).
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 71 | 57
Number analyzed (Attacks requiring Icatibant) | 181 | 453
Attacks requiring Icatibant
  requiring 1 injection | 129 | 306
  requiring 2 injections | 38 | 89
  requiring 3 injections | 13 | 30
  requiring >= 4 injections | 1 | 28

10. Secondary Outcome: Number of Patients With Adverse Events (AEs)
Description: Treatment-emergent adverse events (TEAE) were counted by the treatment most recently taken when the event occurred. Participants were counted once per category per treatment.
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 71 | 57
Participants
  Any TEAE | 42 | 32
  Serious TEAE | 2 | 3
  Severe TEAE | 4 | 3
  TEAE within 24 hours of IP administration | 10 | 7
  Serious TEAE within 24 hours of IP administration | 0 | 0
  Treatment-related TEAE within 24 hrs of IP admin. | 3 | 2
  Treatment-related SAE within 24 hrs of IP admin. | 0 | 0
  TEAE within 24 hrs IP admin. leading to withdrawal | 1 | 0
  Deaths due to TEAE | 0 | 0
  Hospitalizations due to TEAE | 2 | 3
  TEAE leading to withdrawal | 1 | 2
  Treatment-related TEAE | 5 | 4
  Treatment-related SAE | 0 | 0
  Treatment-related severe TEAE | 0 | 0
  Treatment-related TEAE leading to withdrawal | 1 | 0

11. Secondary Outcome: Number of Participants With Injection Site Reactions
Description: Injection site reactions (Erythema, Swelling, Cutaneous pain, Burning sensation, Itching/Pruritus, Warm sensation) were recorded on a designated eCRF page by the site personnel who monitored the local reaction for 1 hour after IP administration 5 times during each treatment period.
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 71 | 57
Participants
  Any injection site reaction | 42 | 15
  Any severe injection site reaction | 2 | 0
  Any mild injection site reaction | 42 | 15
  Any moderate injection site reaction | 14 | 1

12. Secondary Outcome: Number of Patients With Positive Anti-C1 INH Antibodies
Description: Anti-C1 INH antibodies were measured during study time.
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 71 | 57
Participants
  Positive anti-C1 INH antibodies prior treatment | 0 | 0
  Positive anti-C1 INH antibodies developed | 0 | 0

13. Secondary Outcome: PK Parameters: AUC (0-96) and AUC (0-t) for Functional C1 INH Binding Activity
Description: AUC(0-96)=area under the plasma concentration-time curve from time zero to last measurable concentration; AUC(0-t)=area under the plasma concentration-time curve from time zero extrapolated to the end of the dosing interval tau, where tau is approximately 84 hours (ie, average of every 3 or 4 days) AUC(0-96) = AUC(0-tau).
Time Frame: Within 15 min prior dosing at week 1, week 2, week 8, week 16, week 24, week 27/28 and 48 (± 3) hours after dose in week 27/28 in period 1 and 2. In addition 24 (±3) hours, 72 (±6) hours and 96 (±6) hours post dose in week 28 for period 2.
Population: All participants included who have taken at least one dose of investigational product and for whom the primary PK data are considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: mU*h/mL
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 6 | 3
mU*h/mL
  AUC (0-96) | 31070 (17396) | 13860 (7269.0)
  AUC (0-t) | 31190 (17389) | 13860 (7268.3)

14. Secondary Outcome: PK Parameters: AUC (0-96) and AUC (0-t) for C1 INH Antigen Concentrations
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 6 | 3
mcg*h/mL
  AUC (0-96) | 6882 (4586.0) | 1849 (426.36)
  AUC (0-t) | 6902 (4574.0) | 1849 (426.09)

15. Secondary Outcome: PK Parameters: AUC (0-96) and AUC (0-t) for Complement C4 Concentrations (Treamtment C1 INH)
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Treatment C1 INH
Number analyzed (Participants) | 5
mg*h/L
  AUC (0-96) | 16690 (803.60)
  AUC (0-t) | 16780 (895.63)

16. Secondary Outcome: PK Parameters: AUC (0-96) and AUC (0-t) for Complement C4 Concentrations (Treatment Placebo)
Description: AUC(0-96)=area under the plasma concentration-time curve from time zero to last measurable concentration; AUC(0-t)=area under the plasma concentration-time curve from time zero extrapolated to the end of the dosing interval tau, where tau is approximately 84 hours (ie, average of every 3 or 4 days) AUC(0-96) = AUC(0-tau). Participant wise data was reported for this outcome.
Time Frame: as for outcome 13
Population: All participants included who have taken at least one dose of investigational product and for whom the primary PK data are considered sufficient and interpretable. No summary analysis was done and participant wise data are reported.
Measure: Number; unit: mg*h/L
Arm/Group | Treatment Placebo
Number analyzed (Participants) | 2
mg*h/L
  AUC (0-96) - Participant 1 | 8840
  AUC (0-96) - Participant 2 | 2150
  AUC (0-t) - Participant 1 | 8840
  AUC (0-t) - Participant 2 | 2150

17. Secondary Outcome: PK Parameters: Cmax and Cmin for Functional C1 INH Binding Activity
Description: Cmax=maximum observed plasma concentration and Cmin=minimum observed plasma concentration
Time Frame: Within 15 min prior dosing at week 1, week 2, week 8, week 16, week 24, week 27/28 and 48 (± 3) hours after dose in week 27/28 in period 1 and 2 and in addition 24 (±3) hours, 72 (±6) hours and 96 (±6) hours post dose in week 28 for period 2.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 6 | 3
mU/mL
  Cmax | 396.20 (273.013) | 159.50 (82.982)
  Cmin | 258.15 (138.232) | 125.90 (62.329)

18. Secondary Outcome: PK Parameters: Cmax and Cmin for C1 INH Antigen Concentrations
Description: Cmax=maximum observed plasma concentration and Cmin=minimum observed plasma concentration
Time Frame: as for outcome 17
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 6 | 3
µg/mL
  Cmax | 77.680 (52.4375) | 21.257 (5.1647)
  Cmin | 65.562 (45.9331) | 17.913 (4.4316)

19. Secondary Outcome: PK Parameters: Cmax and Cmin for Complement C4 Concentrations (Treatment C1 INH)
Description: Cmax=maximum observed plasma concentration and Cmin=minimum observed plasma concentration
Time Frame: as for outcome 17
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Treatment C1 INH
Number analyzed (Participants) | 5
mg/L
  Cmax | 200 (30.82)
  Cmin | 158 (13.04)

20. Secondary Outcome: PK Parameters: Cmax and Cmin for Complement C4 Concentrations (Treatment Placebo)
Description: Cmax=maximum observed plasma concentration and Cmin=minimum observed plasma concentration. Participant wise data was reported for this outcome.
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Number; unit: mg/L
Arm/Group | Treatment Placebo
Number analyzed (Participants) | 2
mg/L
  Cmax - Participant 1 | 120
  Cmax - Participant 2 | 27
  Cmin - Participant 1 | 82
  Cmin - Participant 2 | 18

21. Secondary Outcome: PK Parameters: Tmax
Description: tmax=time of maximum observed plasma concentration
Time Frame: as for outcome 17
Population: All participants included who have taken at least one dose of investigational product and for whom the primary PK data are considered sufficient and interpretable. For Complement C4 Concentration no summary analysis was done for participants in the placebo group and participant wise data for 2 participants are reported in Outcome measure #19.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 6 | 3
hours
  Functional C1 INH Binding Activity | 31.597 (12.7038) | 55.689 (49.4851)
  C1 INH Antigen Concentration | 31.656 (24.6912) | 47.578 (47.3106)
  Complement C4 Concentration: number analyzed (Participants) | 5 | 0
  Complement C4 Concentration | 33.417 (36.5183) |

22. Secondary Outcome: PK Parameters: Tmax for Complement C4 Concentrations (Placebo Group)
Description: tmax=time of maximum observed plasma concentration. Participant wise data was reported for this outcome.
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Number; unit: mg/L
Arm/Group | Treatment Placebo
Number analyzed (Participants) | 2
mg/L
  tmax - Participant 1 | 94.62
  tmax - Participant 2 | 48.12

23. Secondary Outcome: Assess Disease Activity as Measured by the Angioedema Activity Score (AAS) Normalized Per Month
Description: Disease activity was measured using a 98-day Angioedema Activity Score (AAS). The AAS collects information of disease activity in the last 24 hours. The following items are assessed: experience of swelling, severity of the swelling, timing of the swelling, extent of discomfort due to the swelling, extent that the swelling caused limitations in daily life, and feelings of being disfigured by the swelling. The instrument uses a binary response option for the first item and a three-point response scale for the 5 items thereafter. The daily AAS was the sum of the AAS items per day. Total daily ASS scores range between 0 and 15 points. Higher values stand for higher disease activity. The normalized 98-day AAS per month for a participant is calculated by (the sum of daily AAS within a treatment period/the number of days that a subject has AAS records within the treatment period)*30.4.
Time Frame: Weeks 1 to 14 for treatment period 1 and 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 56 | 57
Score on a scale | 25.433 [11.204 to 39.662] | 57.168 [43.010 to 71.326]
Statistical Analysis 1: Comparison: Treatment C1 INH vs Treatment Placebo; The Least Square means, 95% confidence intervals and p-values are based on mixed effect linear model with period, sequence, use of prophylactic therapy with C1 INH at randomization and treatment as fixed effects and subject nested within sequence as a random effect; Test type: Other; p = 0.0001, Mixed Models Analysis; Difference in LS means = -31.735, 95% CI 2-sided [-42.696 to -20.773]

24. Secondary Outcome: Participant Experience With Self-administration: Overall Experience With the Syringe
Description: Self-administration survey with questions about the overall experience with the syringe was assessed in week 14 (visit 28 and 28b). Visit 28 summarizes treatment period 1 of the experimental/experimental arm and treatment periods 1 and 2 of the experimental/placebo arm and the placebo/experimental arm. Visit 28b summarizes treatment period 2 of the experimental/experimental arm.
Time Frame: Week 14 for treatment period 1 and 2
Population: Visit 28b summarizes only treatment period 2 of the Experimental/Experimental arm. Therefore no participants were analyzed in the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 59 | 40
Participants
  Visit 28: Easy to use | 48 | 36
  Visit 28: Somewhat difficult to use | 11 | 4
  Visiti 28: Difficult to use | 0 | 0
  Visit 28b: Easy to use: number analyzed (Participants) | 12 | 0
  Visit 28b: Easy to use | 11 |
  Visit 28b: Somewhat difficult to use: number analyzed (Participants) | 12 | 0
  Visit 28b: Somewhat difficult to use | 1 |
  Visiti 28b: Difficult to use: number analyzed (Participants) | 12 | 0
  Visiti 28b: Difficult to use | 0 |

25. Secondary Outcome: Participant Experience With Self-administration: How Many Visits for Confidence With Self-administration
Description: The self-administration survey includes the number of visits needed for participants to be able to self-administer investigational product with confidence and all participants could self-administer without supervision. Visit 28 summarizes treatment period 1 of the experimental/experimental arm and treatment periods 1 and 2 of the experimental/placebo arm and the placebo/experimental arm. Visit 28b summarizes treatment period 2 of the experimental/experimental arm.
Time Frame: Week 14 for treatment period 1 and 2
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 59 | 40
Number of visits
  Visit 28 | 1.8 (1.70) | 2.0 (2.49)
  Visit 28b: number analyzed (Participants) | 12 | 0
  Visit 28b | 1.8 (1.22) |

26. Secondary Outcome: Participant Experience With Self-administration: Better Long-term Option and Preferred Administration
Description: as for outcome 25
Time Frame: Week 14 for treatment period 1 and 2
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment C1 INH | Treatment Placebo
Number analyzed (Participants) | 59 | 40
Participants
  Visit 28: SC better long term option | 57 | 39
  Visit 28: IV better long term option | 2 | 1
  Visit 28: SC preferred administration | 56 | 40
  Visit 28: IV preferred administration | 3 | 0
  Visit 28: Preference for admin - very strong | 47 | 33
  Visit 28: Preference for admin - fairly strong | 12 | 6
  Visit 28: Preference for admin - not very strong | 0 | 1
  Visit 28b: SC better long term option: number analyzed (Participants) | 12 | 0
  Visit 28b: SC better long term option | 12 |
  Visit 28b: IV better long term option: number analyzed (Participants) | 12 | 0
  Visit 28b: IV better long term option | 0 |
  Visit 28b: SC preferred administration: number analyzed (Participants) | 12 | 0
  Visit 28b: SC preferred administration | 11 |
  Visit 28b: IV preferred administration: number analyzed (Participants) | 12 | 0
  Visit 28b: IV preferred administration | 1 |
  Visit 28b: Preference for admin - very strong: number analyzed (Participants) | 12 | 0
  Visit 28b: Preference for admin - very strong | 11 |
  Visit 28b: Preference for admin - fairly strong: number analyzed (Participants) | 12 | 0
  Visit 28b: Preference for admin - fairly strong | 0 |
  Visit 28b: Preference for admin - not very strong: number analyzed (Participants) | 12 | 0
  Visit 28b: Preference for admin - not very strong | 1 |

27. Secondary Outcome: Mean Change in Angioedema Quality of Life Questionnaire Scores From Baseline to Week 13
Description: The AE-QoL is a questionnaire on the quality of life of patients suffering from recurrent angioedema. It consists of 17 specific questions that are associated with work, physical activity, free time, social relations, and food. Each of the 17 questions has a five-point response scale ranging from 1 (Never) to 5 (Very Often). The AE-QoL consists of 4 dimensions (functioning=4 questions(qns) fatigue/mood=5 qns, fears/shame=6 qns, nutrition=2 qns) and a total score (all 17 questions).All scores were calculated by using the following formula: (Σ items - min Σ items / max Σ items - min Σ items) x 100. Σ items=sum of response by participant, min Σ items=minimum response possible, max Σ items=maximum response possible. Scores range from 0 to 100 , with higher scores indicating greater impairment. Absolute change calculated as visit score at week 13 minus score at baseline per period.
Time Frame: Baseline to week 13 for treatment period 1 and 2
Measure: Mean (Standard Deviation); unit: Mean change in AE-QoL scores
Groups:
- Experimental/Placebo Arm - Treatment C1 INH: Participants randomized to the Experimental/Placebo arm received C1 Esterase Inhibitor (C1 INH) in treatment period 1.
- Experimental/Placebo Arm - Treatment Placebo: Participants randomized to the Experimental/Placebo arm received Placebo in treatment period 2.
- Placebo/Experimental Arm - Treatment Placebo: Participants randomized to the Placebo/Experimental arm received Placebo in treatment period 1.
- Placebo/Experimental Arm - Treatment C1 INH: Participants randomized to the Placebo/Experimental arm received C1 Esterase Inhibitor (C1 INH) in treatment period 2.
- Experimental/Experimental Arm - Period 1 Treatment C1 INH: Participants randomized to the Experimental/Experimental arm received C1 Esterase Inhibitor (C1 INH) in treatment period 1.
- Experimental/Experimental Arm - Period 2 Treatment C1 INH: Participants randomized to the Experimental/Experimental arm received C1 Esterase Inhibitor (C1 INH) in treatment period 2.
Arm/Group | Experimental/Placebo Arm - Treatment C1 INH | Experimental/Placebo Arm - Treatment Placebo | Placebo/Experimental Arm - Treatment Placebo | Placebo/Experimental Arm - Treatment C1 INH | Experimental/Experimental Arm - Period 1 Treatment C1 INH | Experimental/Experimental Arm - Period 2 Treatment C1 INH
Number analyzed (Participants) | 31 | 28 | 29 | 25 | 15 | 15
Mean change in AE-QoL scores
  AE-QoL Total | -10.35 (17.75) | 4.77 (12.14) | -6.86 (10.72) | -12.10 (9.83) | -11.65 (9.87) | -0.52 (6.58)
  Functioning | -9.25 (21.29) | 6.11 (20.62) | -10.56 (17.23) | -23.33 (19.45) | -20.50 (14.62) | -2.78 (10.34)
  Fatigue/Mood | -8.40 (21.94) | 2.44 (14.20) | -9.11 (10.16) | -10.10 (13.42) | -8.40 (12.29) | 3.11 (9.33)
  Fear/Shame | -12.50 (21.46) | 5.19 (12.06) | -1.67 (10.62) | -5.40 (10.67) | -9.67 (11.91) | -1.85 (11.19)
  Nutrition | -11.00 (22.45) | 6.67 (19.70) | -9.44 (25.55) | -14.76 (17.50) | -8.00 (16.19) | -1.11 (7.82)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time the informed consent was signed through 7 days afer the last dose of investigational product was received (week 1 to 15 for treatment period 1 and 2).
Arm/Group | Treatment C1 INH | Treatment Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/57
Serious Adverse Events (participants affected / at risk) | 2/71 | 3/57
Other Adverse Events (participants affected / at risk) | 23/71 | 14/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment C1 INH (N=71) | Treatment Placebo (N=57)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Hereditary angioedema (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment C1 INH (N=71) | Treatment Placebo (N=57)
Viral upper respiratory tract infection (Infections and infestations) | 11 (11) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 6 (10) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (6):
  • Study Protocol: Protocol (2015-05-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT02584959/Prot_000.pdf
  • Study Protocol: Amendment1 (2015-07-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT02584959/Prot_001.pdf
  • Study Protocol: Amendment2 (2015-09-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT02584959/Prot_002.pdf
  • Study Protocol: Amendment3 (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02584959/Prot_003.pdf
  • Study Protocol: Amendment4 (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT02584959/Prot_004.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT02584959/SAP_005.pdf